CLINICAL TRIAL: NCT04976621
Title: A Feasibility Study of Behavioral Activation in the Rehabilitation of Veterans With Post-TBI Depression
Brief Title: ACTIVE: Activity Therapy to Increase Veteran Engagement
Acronym: ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3578-P
Record Dates: First submitted 2021-07-01; First posted 2021-07-26 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
Keywords: rehabilitation; depression; veterans
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: At the baseline interview, the interviewer will review the study, answer questions, obtain Informed Consent, conduct screening for eligibility, and conduct the baseline interview. The interview will be conducted in the rehabilitation clinic office, by VA Video Connect, or in the home. Veterans who do not wish to continue with the study after the baseline interview will not be randomized.
  Within 48 hours of the baseline interview, eligible veterans will be randomized using the method of random permuted blocks and concealed allocation. Those randomized to BA will be contacted within 5 days by the interventionist and scheduled for the first session. They will receive the 6-session BA intervention (as well as treatment as usual [TAU]). Control participants will receive TAU only (which may include current medical and mental health treatments.) Three months after Baseline, a blinded interviewer will conduct the follow-up interview in person or on the phone with all veterans.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers at the medical center will not have knowledge of the intervention or control condition assigned to individual participants. The research interviewer at the follow-up interview (the outcome assessor) also has no knowledge of the intervention or control condition assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Activation (BA) intervention group (Experimental): Participants in the BA group will receive BA treatment and treatment as usual. BA is a brief behavioral treatment that helps people define goals, create and execute plans to attain them, and engage in meaningful activities. The BA intervention will be delivered in 6 sessions over 3 months by Occupational Therapists trained in BA for post-TBI depression. BA sessions will be conducted in person in an office at the VA rehabilitation clinic, virtually by VA Video Connect, or in person in the home, depending on the veteran's preference.
  Interventions: Behavioral: Behavioral Activation; Other: Treatment as Usual
- Treatment as Usual Control Group (Other): Participants in the Control group receive treatment as usual (TAU), which is usual care provided by the VA medical center.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioral Activation — BA is a brief behavioral treatment that helps people define goals, create and execute plans to attain them, and engage in meaningful activities. BA protocol components include: goal setting (especially for activities that promote social connectedness), creation of a plan (broken down into steps), strategies for implementation of steps, identification of potential barriers, tactics to overcome them, activity monitoring and scheduling, and emotion regulation strategies. The BA intervention will be delivered in 6 sessions over 3 months by Occupational Therapists trained in BA for post-TBI depression. BA sessions will be conducted in person in an office at the VA rehabilitation clinic, virtually by VA Video Connect, or in person in the home, depending on the veteran's preference.
  Arms: Behavioral Activation (BA) intervention group
Other: Treatment as Usual — Treatment as Usual refers to usual care provided by the VA medical center.

SUMMARY:
Depression is common after traumatic brain injury (TBI) and may have wide-ranging consequences. Post-TBI depression may impede reintegration into the family and community and lead to lower quality of life and heightened suicide risk. It may also interfere with rehabilitation. Yet, current treatments for post-TBI depression are based largely on expert opinion rather than evidence from rigorous studies.

Behavioral activation (BA) is a promising intervention for post-TBI depression. It is a brief behavioral treatment that helps people define goals, create and execute plans to reach them, and engage in meaningful activities. BA has been tested in clinical trials since the 1970s and has been shown to reduce or prevent depression in populations with diverse medical conditions. However, BA has rarely been used or studied for treatment of depression in a TBI population.

The investigators will conduct a study of BA with at least 40 Veterans with TBI and depressive symptoms in VA outpatient rehabilitation care. One group of Veterans will be randomly assigned to receive BA plus usual care. The BA program consists of six sessions delivered over three months at the VA (or Veterans' homes, if preferred) by an occupational therapist (OT). A second group of Veterans will be randomly assigned to receive usual care. The investigators will assess the feasibility of delivering the BA intervention in the rehabilitation setting and its acceptability to Veterans and staff. The research team will also assess participant responses to BA in the outcomes of depressive symptoms, community reintegration, and quality of life. Study findings will be used to guide the development of a future study of BA in a larger sample of Veterans with post-TBI depression.

This study and future research may add a powerful clinical tool to rehabilitation services to lessen or prevent depression in Veterans with TBI. Reducing depression may in turn facilitate rehabilitation and enhance community reintegration, allowing Veterans to engage more fully in their families and communities.

DETAILED DESCRIPTION:
Objectives: Nearly 400,000 Veterans have been diagnosed with traumatic brain injury (TBI) since 2000, representing up to 22% of combat casualties. Depression is one of the most prevalent and serious of TBI sequelae. Post-TBI depression adversely affects rehabilitation, treatment adherence, community reintegration (CR), quality of life (QOL), social relationships, and caregiver burden. Yet, post-TBI depression remains under-assessed, undertreated, and under-studied. No clinical guidelines for post-TBI depression treatment exist, and current treatment is largely based on expert opinion rather than evidence from controlled clinical trials.

A promising therapeutic approach to post-TBI depression is Behavioral Activation (BA), a brief and pragmatic treatment rigorously tested since the 1970s in clinical trials for depression in diverse clinical populations. BA helps individuals set goals, create plans, and engage in activities that improve mood and maintain social connectedness - making it well-suited to treating depression in a TBI population that struggles to set goals and is prone to social isolation. BA can accommodate hallmark deficits of TBI such as deficits in memory, organization, planning, initiation, emotion regulation, and interpersonal functioning. It can be delivered by professionals routinely available in VA outpatient rehabilitation services (e.g., occupational therapists, nurses, psychologists, social workers) and, therefore, can be deployed in rehabilitation settings.

The proposed research will assess the feasibility of a BA protocol adapted for post-TBI depression in an outpatient VA rehabilitation setting. Specific study objectives are to: (1) assess BA's acceptability to Veterans and staff and other feasibility indices, (2) provide preliminary evidence of participant response in the outcomes of depressive symptoms, CR, and QOL at the 3-month follow-up interview, (3) develop the BA protocol and manual to be tested in a larger randomized controlled trial (RCT) in the future, and (4) explore engagement in activity as the mechanism that underlies BA intervention effects on outcomes.

Research Design: This feasibility study includes a pilot randomized controlled trail to examine participant response.

Methodology: This feasibility study will enroll at least 40 male and female Veterans receiving care at a VAMC Rehabilitation Medicine Service and meeting study criteria for TBI and depression. Veterans will be randomly assigned to BA plus treatment as usual (TAU) or control (TAU). The BA program consists of six sessions delivered over 3 months at the VA (or the Veteran's home, as preferred by Veteran) by an occupational therapist (OT). All Veterans are interviewed at baseline before randomization and 3 months later by a blinded interviewer. Both interviews assess Veterans' depressive symptoms, CR, and QOL, using standardized instruments. Feasibility will be assessed in six domains: acceptability to Veterans and clinic staff; process (recruitment, refusal, and retention rates; study completion; eligibility criteria; and number of sessions attended); practicality (resources and constraints imposed by the setting); safety; participant comprehension of interviews and the intervention; and research burden (length of interviews, participant fatigue, and emotional distress). After the follow-up interview, phone interviews with BA participants and with clinic staff will be conducted to capture acceptability and their experience with BA. These qualitative and quantitative methods are designed to test the feasibility of a future RCT, identify the barriers and facilitators to implementation of BA in the rehabilitation setting, and describe Veterans' experiences with BA.

Impact/Significance: This study and line of research has the potential to advance knowledge by identifying a feasible and efficacious approach to preventing and/or mitigating depression among Veterans with TBI, a clinical population at high risk for depression and its sequelae. Findings will be used to inform the development of a future RCT powered to test BA's efficacy in a larger sample of Veterans with post-TBI depression.

ELIGIBILITY:
Inclusion Criteria:

* Veteran enrolled in the outpatient Rehabilitation Medicine Service at the Corporal Michael J. Crescenz VA Medical Center
* Age of 21 years or older
* Meet professional criteria for mild or moderate TBI
* Confirmation of TBI diagnosis
* Have a CES-D score at or above 16 at both the Telephone Screen and Baseline
* Those taking antidepressants or other medications affecting mood or behavior must have been using these for at least three months, to allow for stabilization.
* Those in psychotherapy can participate if therapy has been ongoing for three months or longer.
* Veterans report current TBI-related symptoms on the Telephone Screen.
* Speak English

Exclusion Criteria:

* A diagnosis of severe TBI
* Psychosis
* Aphasia
* History of bipolar disorder
* Presence of suicidal ideation with affirmative response on item 9 of the PHQ-9
* History of severe physical aggressiveness, judged by the clinical team
* Currently receiving Cognitive Behavioral Therapy for depression
* Dementia (determined on case-by-case basis based on physician diagnosis and participant's difficulty understanding interview questions)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helene J Moriarty, PhD RN, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the research will be shared outside VA. A de-identified, anonymized dataset will be created and shared. A final dataset will be made available to the public upon receipt of a study-specific Data Use Agreement made in writing and following IRB and VA R&D regulations. Data will be provided electronically and per VA regulations for transferring data.
Supporting Information: Analytic Code
Time Frame: The IDP will be shared starting six months after the publication.
Access Criteria: We will consult with a VA privacy officer and other regulatory specialists at the Corporal Michael Crescenz VA Medical Center, taking all recommended steps to insure that re-identifying participants from the final de-identified and anonymous dataset will not be possible. In addition, the Data Use Agreement will explicitly prohibit attempts to re-identify participants.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants were consented and enrolled, but 5 were deemed ineligible after the baseline interview (1 with CES-D score < 16; 3 with suicidal ideation on item 9 of the PHQ-9; and 1 with inability to take part in the interview).
Period: Overall Study
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
Started | 19 | 22
Completed | 16 | 19
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.16 (14.61) | 47.32 (11.11) | 47.24 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 13 | 10 | 23
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 22 | 41
Depressive Symptom Scores on CES-D [Mean (Standard Deviation); unit: units on a scale] — Total scores may range from 0 to 60, with higher scores indicating greater depressive symptoms.
  units on a scale | 35.56 (6.45) | 31.58 (6.30) | 33.78 (6.60)
Community Reintegration Scores on PART-O-17 [Mean (Standard Deviation); unit: Z score] — The Participation Assessment with Recombined Tools-Objective scale measures participation in the community in 3 domains: Productivity, Out and About, and Social Relations. In our study, scores were converted to z scores because more than one response format was used across items. When data are converted to z scores, the sample mean is always 0. Scores (i.e., z scores, not standard deviations) above 0 indicate better than average community participation, those below 0 indicate worse participation. Higher scores of this scale indicate better participation.
  Z score | .07 (.34) | -.03 (.30) | -0.00 (.33)
Quality of Life in TBI Scores on QoL-TBI Instrument [Mean (Standard Deviation); unit: units on a scale] — This tool uses a 5-point scale from "0 - Not at all" to "4- Very." Although the published description of this tool designates sums across all items as a summary score, we computed means scores of all items. The reason is that the use of a sum poses a problem whenever there are missing data, which produces a spuriously lower score for individuals with some missing responses. Higher scores indicate better quality of life.
  units on a scale | 1.90 (.31) | 2.00 (.40) | 1.94 (.36)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Scores on CES-D
Description: Depressive symptoms will be measured by The Center for Epidemiologic Studies Depression Scale (CES-D). CES-D is a well-established 20-item screening instrument that shows good psychometric properties in TBI populations. It will be administered at the Baseline interview and Follow-up interview (at 3 months). It uses a Likert-type scale from 0 to 3. The total score is the sum across all 20 items. Total scores may range from 0 to 60, with higher scores indicating greater depressive symptoms.
Time Frame: 3 - 4 months
Population: Forty-six Veterans were enrolled. After consenting and the baseline interview, 5 were deemed ineligible for the study. Therefore, 41 Veterans were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 16 | 19
units on a scale | 30.06 (9.30) | 29.68 (11.70)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group vs Treatment as Usual Control Group; This feasibility study assessed preliminary evidence of treatment response. We have reported only descriptive statistics for quantitative findings. We have not reported inferential statistics, in keeping with the purpose of the VA SPiRE grant mechanism through which the study was funded. We assessed change in participant response by comparing the mean change in the outcome from baseline to follow-up in Group 1 (BA) and Group 2 (TAU). We inspected trends and directions of change in both groups; Test type: Other — Because this was a feasibility study, we did not compute inferential statistics and did not include a power calculation; Because this was a feasibility study, inferential statistics were not computed; Because this is a feasibility study, inferential statistics were not computed. We examined the trends and direction of change in the baseline mean score and follow-up mean score between the two groups

2. Secondary Outcome: Community Reintegration Scores on PART-O-17
Description: The Participation Assessment with Recombined Tools-Objective scale (PART-O-17) measures participation in the community in three domains: Productivity, Out and About, and Social Relations. In our study, scores were converted to z scores because more than one response format was used across items. When data are converted to Z scores, the sample mean is always 0. Scores (i.e., Z scores, not standard deviations) above 0 indicate better than average community participation, those below 0 indicate worse participation. Thus, higher scores of this scale indicate better participation.
Time Frame: 3 - 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 16 | 19
Z score | .13 (.38) | -.11 (.23)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group vs Treatment as Usual Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Quality of Life in TBI Scores on QoL-TBI Instrument
Description: Quality of life in TBI will be measured by The QoL-TBI instrument. This is a 37-item patient-centered measure that captures the individual's perception of his/her health-related quality-of-life (HRQoL) in cognition, self-care, daily life and autonomy, social relationships, emotions, and physical problems. It will be administered at the Baseline interview and Follow-up interview (at 3 months). It uses a 5-point scale from "0 - Not at all" to "4- Very." Although the published description of this tool designates sums across all items as a summary score, we computed the mean of all items. The reason is that the use of a sum poses a problem whenever there are missing data, which produces a spuriously lower score for individuals with some missing responses. Higher scores indicate better quality of life.
Time Frame: 3 - 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 16 | 19
units on a scale | 2.05 (.47) | 1.92 (.40)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group vs Treatment as Usual Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Other Pre Specified Outcome: Acceptability of the Intervention Rated by the Interventionist
Description: Acceptability is measured by the Acceptance/Receipt Scale and is completed by the interventionist at the last intervention session. This is an 18-item tool with Likert scale response formats from 0 to 4. A mean score will be obtained and ranges from 0 to 4. Higher scores indicate increased acceptability.
Time Frame: 3 - 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) Intervention Group
Number analyzed (Participants) | 14
units on a scale | 2.75 (.36)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group; Test type: Other; Descriptive statistics are being used

5. Other Pre Specified Outcome: Veteran Acceptability/Satisfaction With the Intervention
Description: Acceptability/Satisfaction with the intervention will be measured with the Acceptability/Satisfaction Scale and is completed by the participants who received Behavioral Activation after the last intervention session when the qualitative interview is also conducted. This is a 12 item tool with a Likert scale response format from 0 to 4. A mean score will be obtained and ranges from 0 to 4. A higher score indicates increased acceptability/satisfaction.
Time Frame: 3 - 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) Intervention Group
Number analyzed (Participants) | 5
units on a scale | 3.34 (1.59)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group; Descriptive statistics are used to describe acceptability/satisfaction for those who received the BA intervention. This tool is completed after the last intervention session when the qualitative interview is also conducted; Test type: Other; Descriptive statistics are used in this feasibility study. We are not using inferential statistics to test for statistical significance

6. Other Pre Specified Outcome: Recruitment
Description: Recruitment is considered part of the process domain of feasibility. Recruitment will be measured by the percentage of veterans eligible for the study among those screened and the percentage willing to participate among those screened. Among those screened, our criteria for recruitment is that 50% or more will be eligible for the study and that at least 30% will be willing to participate.
Time Frame: 16 months
Population: This is the total number who completed the initial telephone screen. This involved screening for all potential participants prior to randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation (BA) Intervention Group
Number analyzed (Participants) | 72
Participants
  Not eligible | 6
  Consented | 46
  Refused to participate | 20
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group; Test type: Other; Descriptive statistics are used to describe recruitment

7. Other Pre Specified Outcome: Retention
Description: Retention is considered part of the process domain of feasibility and will be measured in two ways. Retention will be measured by the number of treatment sessions completed over the total number of sessions (6) for only those in the treatment group. The percentage who completed at least four treatment sessions will be the criterion for this. Among those who are enrolled in both groups, retention is measured by the percentage in each group who completed the Time 2 follow-up interview (which occurred 3 - 4 months after the baseline interview).
Time Frame: 3 - 4 months for the number in each group that completed the Time 2 follow-up interview and up to 4 months for number in treatment group who completed at least four treatment sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 19 | 22
Participants
  Retention - Number in each group that completed the Time 2 follow-up interview | 16 | 19
  Retention - Number in treatment group who completed at least four treatment sessions | 16 | 0
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group vs Treatment as Usual Control Group; Test type: Other; One measure of retention was the percent in each group who completed the study, meaning completed the Time 2 follow-up interview (that occurred 3-4 months after the baseline interview). Another measure of retention was the percent in the treatment group that completed four or more treatment sessions

8. Other Pre Specified Outcome: Treatment Fidelity
Description: Treatment fidelity is considered part of the process domain of feasibility. This will be measured by the Treatment Fidelity Checklist, a 15-item tool with a 3-point scale with responses from 1 (poor) to 3 (excellent). The mean will be computed for the 15 items for each recorded interview. The percentage of the interviews that had a mean less than 2.0 will be computed and will be the measure of treatment fidelity. Our criterion is that no more than 15% of sessions observed or audiotaped will have a mean less than 2.0.
Time Frame: 18 months
Population: One transcript of a treatment session for each of 5 participants who received treatment was analyzed. Thus, 5 transcripts were analyzed.
Measure: Number; unit: number of transcripts with mean < 2.0
Units Other Than Participants: 5 transcripts of treatment sessions
Arm/Group | Behavioral Activation (BA) Intervention Group
Number analyzed (Participants) | 5
Number analyzed (5 transcripts of treatment sessions) | 5
number of transcripts with mean < 2.0 | 5
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Intervention Group; Test type: Other; For each of five participants who received the intervention, we reviewed a transcript of 1 intervention session for treatment fidelity. The criterion is that no more than 15% of sessions observed or audiotaped will have a mean less than 2.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent until the final study contact, up to 21 months.
Arm/Group | Behavioral Activation (BA) Intervention Group | Treatment as Usual Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/22
Other Adverse Events (participants affected / at risk) | 7/19 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (BA) Intervention Group (N=19) | Treatment as Usual Control Group (N=22)
Breathing difficulty, diagnosis of acute COPD exacerbation, hospitalized (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Injuries from fall (fractured ribs, concussion, and difficulty with hip and ambulation) (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (BA) Intervention Group (N=19) | Treatment as Usual Control Group (N=22)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
puncture wound of foot (stepped on nail) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COVID 19 (Infections and infestations) | 1 (1) | 0 (0)
strained back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
vertigo flare (Ear and labyrinth disorders) | 1 (1) | 0 (0)
acute cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cut hand requiring 3 stitches (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
neck and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
migraine (Nervous system disorders) | 1 (1) | 0 (0)
deviated septum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
non-specific cold symptoms (General disorders) | 1 (1) | 0 (0)
abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT04976621/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT04976621/ICF_000.pdf